CLINICAL TRIAL: NCT06973837
Title: Unravelling the Neurobiological Mechanisms Underlying the Bidirectional Relationship Between Chronic Sleep Disturbances and Pain Sensitivity in People With Non-specific Chronic Low Back Pain and Chronic Insomnia
Brief Title: Studying the Neurobiological Mechanisms of Non-specific Chronic Low Back Pain and Chronic Insomnia: a Four-group Cross-sectional Study
Acronym: SY-NAPS-CS
Status: Recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Iris Coppieters, Dr. Iris Coppieters (Principal investigator), Vrije Universiteit Brussel
Other Study IDs: 11PMF24N; G080423N (Other Grant/Funding Number: Research Foundation - Flanders); S68780 (Other: Ethics Committee Research UZ/KU Leuven)
Record Dates: First submitted 2025-05-05; First posted 2025-05-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain (CLBP); Chronic Insomnia; Neuroinflammation
Keywords: Pain; Chronic pain; Chronic low back pain; Sleep; Insomnia; Chronic insomnia; Magnetic resonance imaging; Functional magnetic resonance imaging; Magnetic resonance spectroscopy; Diffusion weighted imaging; Quantitative sensory testing; Temporal summation; Conditioned pain modulation; Experience sampling method; Ecological momentary assessment; Microbiota; Gut-Brain axis; Short-chain fatty acids
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neuroinflammatory Diseases; Pain; Chronic Pain | interventions — Neuroimaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Systemic venous blood samples will be taken, from which designated serum will be extracted for the analysis of short chain fatty acids and highly-sensitive C-reactive protein.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pain-free with good sleep habits (healthy controls): Meeting all General inclusion/exclusion criteria and Pharmacological exceptions criteria, plus the specific inclusion criteria for "pain-free" and "good sleeper".
  Interventions: Other: Real-life monitoring, experimental pain testing, brain imaging, blood and stool sampling.
- Non-specific chronic low back pain with good sleep habits: Meeting all General inclusion/exclusion criteria and Pharmacological exceptions criteria, plus the specific inclusion criteria for "chronic low back pain" and "good sleeper".
  Interventions: Other: Real-life monitoring, experimental pain testing, brain imaging, blood and stool sampling.
- Pain-free with chronic insomnia: Meeting General inclusion/exclusion criteria and Pharmacological exceptions criteria, plus the specific inclusion criteria for "pain-free" and "chronic insomnia".
  Interventions: Other: Real-life monitoring, experimental pain testing, brain imaging, blood and stool sampling.
- Non-specific chronic low back pain with comorbid chronic insomnia: Meeting all General inclusion/exclusion criteria and Pharmacological exceptions criteria, plus the specific inclusion criteria for "chronic low back pain" and "chronic insomnia".
  Interventions: Other: Real-life monitoring, experimental pain testing, brain imaging, blood and stool sampling.

INTERVENTIONS:
Other: Real-life monitoring, experimental pain testing, brain imaging, blood and stool sampling. — See detailed study description and outcome measures.

SUMMARY:
This study is a part of a larger project aiming to evaluate the neurobiological mechanisms underlying the relationship between sleep and pain in people with non-specific chronic low back pain. Specifically, this study aims to evaluate the neurobiological mechanisms underlying the relationship between chronic sleep disturbances and pain sensitivity in people with non-specific chronic low back pain and chronic insomnia.

DETAILED DESCRIPTION:
Sleep disturbances, and especially insomnia, reflect one of the most common comorbidities in people with chronic pain, including people with chronic low back pain. Previous research has furthermore demonstrated that a lack of sleep is associated with an increased pain sensitivity. The goal of this study is to evaluate the role of brain neuroinflammation in the relationship between chronic sleep disturbances and both clinical and experimental pain sensitivity in people non-specific chronic low back pain and/or chronic insomnia.

A cross-sectional study will be conducted across four age- and sex-matched study groups: healthy controls with good sleep habits (Group 1); people with non-specific chronic low back pain and good sleep habits (Group 2); pain-free individuals with chronic insomnia (Group 3); and people with non-specific chronic low back pain and comorbid chronic insomnia (Group 4). The study will be performed over nine consecutive days. All participants will arrive at the lab at a standardized time, relative to their habitual bedtime, in the afternoon of the first study day. There, they will first fill out a number of baseline questionnaires, after which a battery of quantitative sensory test, utilizing both manual and computerized pressure algometry, will be performed to assess experimental pain sensitivity. After being provided a standardized dinner, the participants will then perform a clinical polysomnography (i.e., sleep study) during an over-night stay at the hospital sleep center (UZ Leuven, Belgium) to acquire data on sleep time, stability, and efficiency, as well as to identify participants with combined sleep-disorder-comorbidity profiles (e.g. insomnia + apnea). Directly upon awakening in the morning of the second day, all participants will first fill in a few additional questionnaires, and then be provided a standardized low-fiber breakfast alongside a bolus of pure fiber. Next, the participants will be escorted to the magnetic resonance imaging facility and perform two blocks of brain scanning separated by an approximate 10-min break. During the first block, magnetic resonance spectroscopy and diffusion-weighted magnetic resonance imaging will be performed to measure markers of neuroinflammation, whereas the second block utilizes functional magnetic resonance imaging during an evoked-low-back-pain task to acquire data on back pain-evoked brain activity. After the two scanning blocks, the second study day ends by the collection of a venous blood sample to assess systemic levels of inflammation (via highly sensitive C-reactive protein) and short chain fatty acids. During the following seven days, all participants will complete a sleep diary once per day, provide momentary ratings of pain, sleepiness, fatigue, and affect eight times per day, and wear an Actigraph at all times (except during heavy water contact). During this seven-day period, the participants will also be instructed to collect a stool sample at a time of their own convenience, but preferably within the first three days, to be used for gut microbiota composition analyses. Continuous dietary intake will therefore also be recorded during the first three days of the seven-day period, while participants who are not able to collect their stool sample during any of these three days will continue to record their dietary intake until a stool sample has been collected.

ELIGIBILITY:
General inclusion criteria (all groups):

* 18-60 years old.
* Ability to speak and understand the Dutch Language.
* Body mass index <30.
* No smoking or nicotine use.
* Low caffeine use (≤3 cups of coffee/day, ≤1 energy drink/day).
* Low alcohol use (≤9 alcoholic units/week).
* No use of neuro- and/or psychopharmacological treatments and/or immunosuppressive agents (including NSAIDs) with a suspected influence on neuroinflammation unless terminated within a sufficient time frame before the start of the study, or unless falling under the Pharmacological exceptions criteria (see below).
* Willing to (try to) adhere to the acute pre-test restrictions, including refraining from analgesics (unless stable use), caffeine, alcohol, and/or strenuous physical activity (>3 METs) in the 24 hours preceding the main test day.

General exclusion criteria (all groups):

* Shift worker.
* Use of blood thinners.
* (History of) Substance dependence/abuse.
* Chronic pain conditions (≥3 months) other than chronic low back pain.
* Severe intrinsic sleep disorders (assessed during a one-night, laboratory-based polysomnography).
* Restless leg syndrome
* Central or peripheral neurological disorder/condition (e.g., epilepsy, multiple sclerosis, peripheral neuropathy).
* History of spinal surgery.
* Major medical (e.g., cardiac disease, cancer) and/or psychiatric disorder/disease (e.g., major depressive disorder, bipolar disorder).
* Claustrophobia.
* Contraindications for magnetic resonance imaging (e.g., metal/cochlear implants, pacemaker).
* Pregnancy or being <12 months post-natal.

Pharmacological exceptions criteria:

- Participants with chronic low back pain and/or (comorbid) insomnia will be allowed to be on a stable low dose of weak pain and/or sleep agents (e.g., Tramadol, Zolpidem) if medically prescribed specifically for their low back pain and/or insomnia, and if approved by the national medicine register of Belgium (FAMHP, Federal Agency for Medicine and Health Products). These participants will also be allowed stable and/or occasional use of low-to-moderate doses of over-the-counter medications for pain and/or sleep that are suspected to have no or minimal impact on neuroinflammation (e.g., paracetamol, melatonin). Habitual use of medications according to the above-stated criteria should be maintained across the entire study period, with the only exception being analgesics taken on an occasional basis. Specifically, because of the extensive battery of pain tests that will be utilized in the study, all analgesics that are only taken occasionally should be refrained from during the 24 hours preceding the main test day (pre-test instructions).

Specific inclusion criteria for "pain-free" groups:

* Currently pain free, defined as having no pain that affects daily living/functioning and/or which has led to a consultation with a healthcare practitioner.
* No episode of low back pain that interfered with daily functioning/living and/or which led to a consultation with a healthcare practitioner within 12 months from the time of inclusion.
* No history of chronic low back pain.

Specific inclusion criteria for "chronic low back pain" groups:

* Low back pain reported on most days (≥50%), every week, for more than 3 months.
* Low back pain-related emotional disress OR functional disability rated as ≥3 out of 10.

Specific inclusion criteria for "good sleeper" groups:

* Stable sleep phase within 10 PM and 10 AM (assessed using the Pittsburgh Sleep Quality Index).
* Average habitual total sleep time between 7 and 9 hours (assessed using the Pittsburgh Sleep Quality Index).
* A Pittsburgh Sleep Quality Index ≤5.
* An Insomnia Severity Index ≤7.
* An Epworth Sleepiness Scale ≤10.
* Sleep efficiency ≥85% during a one-night, laboratory-based polysomnography screening.
* No episode of sleep disturbances that interfered with daily functioning/living and/or which led to a consultation with a healthcare practitioner within the preceding 12 months from the time of inclusion.
* No history of chronic insomnia.

Specific inclusion criteria for "chronic insomnia" groups:

* Chronic insomnia according to the ICSD-3-TR criteria (assessed using an ICSD-3-TR-adapted version of the Pittsburgh Sleep Quality Index).
* An Insomnia Severity Index ≥15.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants across all study groups will be recruited from the broad area around Leuven, Belgium, via local flyers and social media. Participants with non-specific chronic low back pain and/or chronic insomnia will also be recruited from the pain and/or sleep center of UZ Leuven, Belgium, as well as via primary care units and patient support groups targeting people in the Leuven area. Participants will be recruited and stratified according to sex and age to enable matching to the primary group of interest (chronic low back pain and comorbid insomnia), and a majority of females (~two thirds) will be recruited to better represent the sex-distribution within the population representative of this group.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Brain metabolite concentrations | Day 2
  Concentration of brain metabolites measured using single-voxel magnetic resonance spectroscopy in five regions of interest: (1) pregenual anterior cingulate cortex (midline); (2/3) right/left thalamus; (4/5) right/left anterior insula.

SECONDARY OUTCOMES:
Brain-tissue microstructure diffusivity | Day 2
  Diffusivity data (diffusion-weighted signal) from different microstructural compartments within the brain (intra-axonal space, extra-axonal space, and free water) measured using diffusion-weighted magnetic resonance imaging.
Functional brain responses to evoked low back pain | Day 2
  Blood-oxygen-level-dependent (BOLD) signal acquired during an evoked low back pain task performed during functional magnetic resonance imaging sequence.
Manual pressure pain detection thresholds (mPDT) | Day 1
  Gradually increasing pressure (1 kgf/sec) applied using a manual pressure algometer (FPX50, Wagner Instruments, USA) until the first sensation of discomfort (mPDT) is (self-)reported. The measurement is repeated three times across six body sites: (1/2) right/left m. erector spinae; (3/4) right/left m. extensor carpi radialis; (5/6) right/left m. gastrocnemius.
Computerized pressure pain detection thresholds (cPDT) | Day 1
  Gradually increasing pressure (1 kPa/sec) applied via a computer-controlled blood pressure cuff (Nocitech, Aalborg University, Denmark) around the calf (dominant leg) until a first sensation of discomfort (cPDT) is rated.
Computerized pressure pain tolerance thresholds (cPTT) | Day 1
  Gradually increasing pressure (1 kPa/sec) applied via a computer-controlled blood pressure cuff (Nocitech, Aalborg University, Denmark) around the calf (dominant leg) until it is no longer tolerable.
Temporal summation of (pressure) pain | Day 1
  Twelve repeated pressure stimuli (stimulus duration: 1 sec; interstimulus interval: 1 sec) applied via a computer-controlled blood pressure cuff (Nocitech, Aalborg University, Denmark) around the calf (dominant leg) at an intensity corresponding to the cPTT.
Conditioned (pressure) pain modulation | Day 1
  One cPTT assessment via computer-controlled blood pressure cuff algometry (Nocitech, Aalborg University, Denmark) performed immediately before and after a 1-min hot water immersion of the hand contralateral to the stimulated calf (dominant leg).
Daily self-reported pain distribution assessed via experience sampling methodology (m-Path smartphone application) | Day 3 to 9
  A list of body regions from which participants select the regions at which they experience pain "right now", assessed at eight block-randomized time points per day.
Daily self-reported low back pain (fluctuations) assessed via experience sampling methodology (m-Path smartphone application) | Day 3 to 9
  Intensity, unpleasantness, and attention to low back pain "right now" rated on a 0-to-100 visual analogue scale at eight block-randomized time points per day.
Daily self-reported affect (fluctuations) assessed via experience sampling methodology (m-Path smartphone application) | Day 3 to 9
  Positive and negative affect "right now" rated on a 0-to-100 visual analogue scale at eight block-randomized time points per day.
Daily self-reported fatigue (fluctuations) assessed via experience sampling methodology (m-Path smartphone application) | Day 3 to 9
  Mental and physical fatigue "right now" rated on a 0-to-100 visual analogue scale at eight block-randomized time points per day.
Daily self-reported sleepiness (fluctuations) assessed via the Karolinska Sleepiness Scale (KSS) implemented into the experience sampling methodology smartphone application (m-Path) | Day 3 to 9
  The KSS is a single-item questionnaire (i.e., scale) that measures subjective sleepiness at a specific moment in time. Scores range from 1 to 9, with higher scores indicating greater sleepiness. The scale was completed at eight block-randomized time points per day.
Daily sleep-wake cycles assessed by Actigraphy | Day 3 to 9
  Wrist-worn actigraphy (GT3X Actigraph, Pensacola, FL, USA) at all times except heavy water contact.
Daily self-reported perceived sleep duration assessed via sleep diaries | Day 3 to 9
  Subjective time points for when getting into and out of bed, and for sleep onset and offset, provided once per day.
Daily self-reported nighttime pain assessed via sleep diaries | Day 3 to 9
  Pain intensity during the preceding night, rated on a 0-to-10 numerical rating scale once per day.
Daily self-reported subjective sleep quality assessed via sleep diaries | Day 3 to 9
  Subjective sleep quality from the preceding night, rated on a 0-to-10 numerical rating scale once per day.
Daily self-reported subjective wake quality assessed via sleep diaries | Day 3 to 9
  Subjective wake quality during the day, rated on a 0-to-10 numerical rating scale once per day.
Serum short chain fatty acid levels | Day 2
  Levels of short chain fatty acids analysed from serum aliquots derived from venous blood samples.
Microbiota composition | At one single occasion at any day between Day 3 to 9
  Composition-related outcomes (e.g., diversity, abundance) analysed from stool-sample aliquots.
Habitual self-reported macronutrient intake (including fibre) assessed via continuous dietary records (MyFitnessPal smartphone application) | From Day 3 to at least Day 5, but up to Day 9 depending on the day at which a stool sample is collected
  Macronutrient and fibre intake (in grams) estimated (via MyFitnessPal application) from continuous self-reported dietary intake (food diary).

OTHER OUTCOMES:
Pre-scanning total sleep time | One night between Day 1 and 2
  Polysomnography-derived total sleep time (i.e., min asleep from sleep onset to offset) from the night preceding the brain scanning.
Pre-scanning sleep efficiency | One night between Day 1 and 2
  Polysomnography-derived sleep efficiency from the night preceding the brain scanning.
Self-reported (REDCap) mood state assessed via a short (32-item) version of the Profile of Mood States (POMS-32) | Day 2
  The POMS-32 is a short version of the original 65-item POMS questionnaire, which evaluates mood states across six dimensions: tension-anxiety, depression-dejection, anger-hostility, vigour-activity, fatigue-inertia, and confusion-bewilderment. Total scores for each subscale vary, with higher scores indicating greater intensity of the corresponding mood state.
Self-reported (REDCap) sleepiness assessed via the Karolinska Sleepiness Scale (KSS) | Day 2
  The KSS is a single-item questionnaire (i.e., scale) that measures subjective sleepiness at a specific moment in time. Scores range from 1 to 9, with higher scores indicating greater sleepiness.
Pain distribution assessed via a digital body chart | Day 1 and 2
  A digitalized body chart used to mark all regions at which participants experience pain.
Self-reported (REDCap) pain severity assessed via the Brief Pain Inventory (BPI) | Day 1 and 2
  The BPI is an 11-item questionnaire that evaluates pain severity and the degree to which pain interferes with daily functioning. No total score is obtained, but individual items are rated on 0-to-10 numeric rating scales, with higher ratings indicating greater pain severity or interference.
Self-reported (REDCap) fatigue assessed via the Brugmann Fatigue Scale (BFS) | Day 1
  The BFS is a 10-item questionnaire that evaluates physical and mental fatigue symptoms. Total scores range from 0 to 40, with higher scores indicating greater fatigue severity.
Self-reported (REDCap) sleepiness assessed via the Epworth Sleepiness Scale (ESS) | Day 1
  The ESS is an 8-item questionnaire that evaluates daytime sleepiness by assessing the likelihood of dozing off in various situations. Total scores range from 0 to 24, with higher scores indicating greater daytime sleepiness.
Self-reported (REDCap) morningness/eveningness phenotype assessed via the Morning-Eveningness Questionnaire (MEQ) | Day 1
  The MEQ is a 19-item questionnaire that evaluates an individual's circadian preference by examining preferred times for activities and alertness. Total scores range from 16 to 86, with higher scores indicating a morning preference and lower scores indicating an evening preference.
Self-reported (REDCap) pain hypervigilance assessed via the Pain Vigilance and Awareness Questionnaire (PVAQ) | Day 1
  The PVAQ is a 16-item questionnaire that evaluates the degree of attention individuals pay to pain. Total scores range from 0 to 80, with higher scores reflecting greater pain vigilance and awareness.
Self-reported (REDCap) pain catastrophizing assessed via the Pain Catastrophizing Scale (PCS) | Day 1
  The PCS is a 13-item questionnaire that evaluates catastrophic thinking related to pain, including rumination, magnification, and helplessness. Total scores range from 0 to 52, with higher scores indicating greater pain catastrophizing.
Self-reported (REDCap) pain-related disability assessed via Oswestry Low Back Pain Disability Questionnaire (ODI) | Day 1
  The ODI is a 10-item questionnaire that evaluates the degree of disability related to low back pain across various daily activities. Total scores range from 0 to 100, with higher scores indicating greater disability.
Self-reported (REDCap) insomnia severity assessed via the Insomnia Severity Index (ISI) | Day 1
  The ISI is a 7-item questionnaire that evaluates the nature, severity, and impact of insomnia. Total scores range from 0 to 28, with higher scores indicating more severe insomnia symptoms.
Self-reported (REDCap) sleepiness-related disability assessed via the short (10-item) version of the Functional Outcomes of Sleep Questionnaire (FOSQ-10) | Day 1
  The FOSQ-10 is validated short version of the original FOSQ questionnaire, which evaluates the impact of excessive sleepiness on daily functioning across multiple domains. Total scores range from 5 to 20, with lower scores indicating greater impact on daily functioning due to sleepiness.
Self-reported (REDCap) affect trait assessed via Positive and Negative Affect Schedule (PANAS) | Day 1
  The PANAS is a 20-item questionnaire that evaluates positive and negative affect, with 10 items for each dimension. Total scores range from 10 to 50 for each subscale, with higher scores indicating greater levels of positive or negative affect, respectively.
Self-reported (REDCap) features of depression assessed via the Patient Health Questionnaire-9 (PHQ-9) | Day 1
  The PHQ-9 is a 9-item questionnaire that evaluates the severity of depressive symptoms. Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Self-reported (REDCap) features of anxiety assessed via the General Anxiety Disorder-7 (GAD-7) | Day 1
  The GAD-7 is a 7-item questionnaire that evaluates the severity of generalised anxiety symptoms. Total scores range from 0 to 21, with higher scores indicating greater anxiety severity.
Self-reported (REDCap) stress assessed via the Perceived Stress Scale (PSS) | Day 1
  The PSS is a 10-item questionnaire that measures the degree to which individuals perceive situations in their life as stressful. Total scores range from 0 to 40, with higher scores indicating greater perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ/KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in a publication will be made available to other researchers with all identifying information removed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon publication with no time limitations.
Access Criteria: The data will be publicly available.